CLINICAL TRIAL: NCT04525521
Title: Hand Sanitizer Effects on the Skin Barrier
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS 0720; 3030005053 (Other Grant/Funding Number: National Jewish Health)
Record Dates: First submitted 2020-08-18; First posted 2020-08-25 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Dermatitis Hand; Skin Abnormalities; Atopic Dermatitis; Atopic Dermatitis Eczema
Keywords: Hand dermatitis; Skin barrier; Hand washing; Hand sanitizer; Eczema; Atopic dermatitis
MeSH Terms: conditions — Skin Abnormalities; Dermatitis, Atopic; Eczema | interventions — Hand Sanitizers; Hand Disinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin tape strips will be analyzed for lipid, proteins, and filaggrin breakdown products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Atopic Individuals: Individuals with no history of atopic dermatitis, food allergy, asthma, or allergic rhinitis will be recruited to this cohort. Skin studies (transepidermal water loss and skin tape strips) will be performed on the non-dominant hand at baseline, after hand sanitizer use, and after hand washing with soap and water.
  Interventions: Other: Hand sanitizer and hand washing
- Individuals with Atopic Dermatitis: Individuals with history of atopic dermatitis will be recruited to this cohort. Skin studies (transepidermal water loss and skin tape strips) will be performed on the non-dominant hand at baseline, after hand sanitizer use, and after hand washing with soap and water.
  Interventions: Other: Hand sanitizer and hand washing

INTERVENTIONS:
Other: Hand sanitizer and hand washing — All subjects will cleanse their hands with hand sanitizer, followed by hand washing with soap and water

SUMMARY:
Hand washing and the use of hand sanitizers are important interventions in disease prevention. Engaging in frequent hand washing is especially effective in preventing the spread of viruses, as this removes microbes and prevents the spread to others. Hand dermatitis, however, is a common occurrence in certain occupations, such as healthcare workers. With the onset of the SARS-CoV2 (COVID-19) pandemic, hand hygiene measures are further enforced as there is no cure or vaccine for this virus.

In the study, the effects of hand washing and the use of hand sanitizer on skin proteins and lipids will be assessed.

DETAILED DESCRIPTION:
Hand washing and the use of hand sanitizers are important interventions in disease prevention. Engaging in frequent hand washing is especially effective in preventing the spread of viruses, as this removes microbes and prevents the spread to others. Hand dermatitis, however, is a common occurrence in certain occupations, such as healthcare workers. With the onset of the SARS-CoV2 (COVID-19) pandemic, hand hygiene measures are further enforced as there is no cure or vaccine for this virus.

The stratum corneum is in the outer layer of the epidermis, and it contains several proteins and lipids that are important for skin health. This skin layer can be disrupted by agents that cause skin dryness and irritation, resulting in a dysfunctional skin barrier when there is loss of filaggrin breakdown products, also referred to as natural moisturizing factor (NMF), and lipids. This then leads to the unwanted dermatologic effects of skin dermatitis, and in some patients, contact dermatitis. While it is known that frequent hand washing and hand sanitizer use causes hand dermatitis, the effects on skin barrier proteins and lipids has not been studied.

In this study, the effects of hand washing and the use of hand sanitizer on epidermal proteins and lipids will be assessed. The skin barrier will be examined with skin tape strips (STS) and transepidermal water loss (TEWL) before and after topical skin exposure to hand sanitizer use and hand washing. Questionnaires will be administered to inquire about allergy history, frequency of hand washing, and use of detergents and soaps.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the AD group:

• Individuals with atopic dermatitis, ages 18-60 years old.

Inclusion criteria of the non-atopic group, ages 18-60 years old:

• Individuals with no history of atopic dermatitis, contact dermatitis, food allergy, asthma, or allergic rhinitis.

Exclusion Criteria:

Exclusion criteria of all subjects:

* Subject has taken systemic immunosuppressive drugs including oral steroids within 30 days of skin barrier assessment
* Subject has received immunotherapy in the past year
* Subject has received any biologic medications within 5 half-lives or 16 weeks, whichever is longer
* Subject has received any investigational drugs within 5 half-lives or 8 weeks, whichever is longer
* Subject has taken anti-anxiety, antidepressant, or anticoagulant medications in the last 30 days
* Subject has received total body phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA], tanning beds [>1 visit per week]) within 30 days of skin barrier assessment
* Subject has used topical corticosteroids, topical immunomodulatory agents, or topical antibiotics on the extremity being evaluated within 7 days of skin barrier assessment
* Subject has a severe concurrent disease or immunosuppression
* Subject has a history of a severe reaction to latex, tape, or adhesives
* Subject is pregnant or lactating

For the medications below, they have to be temporarily withheld before participation in the study:

* If the subject is taking oral antihistamines, they will need to be withheld for five days prior to the skin barrier study.
* If the subject is taking oral antibiotics, antivirals, antifungals, or antiparasitics, the skin barrier studies can be scheduled seven days after the last dose has been taken.
* If the subject is taking topical medications including (but not restricted to) Elidel, Protopic, topical corticosteroids and topical antibiotics, they will need to be withheld on the hand being evaluated seven days prior to the skin barrier studies. Moisturizers will also need to be withheld on the area 24 hours prior to the visit. The subject cannot have taken a bleach bath within 7 days of the visit, and the subject cannot take a bath or shower on the day of the visit.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Subjects will have either atopic dermatitis or no history of atopic conditions.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
Measure the change in transepidermal water loss and skin components after using hand sanitizer. | Through study completion, up to 1 year
  Skin barrier assessments at baseline, then after hand sanitizer use will be performed. Analysis of skin filaggrin breakdown products, lipid profiles, and transepidermal water loss will be compared.
Measure the change in transepidermal water loss and skin components after hand washing with soap and water. | Through study completion, up to 1 year
  Skin barrier assessments after hand washing with soap and water will be performed. Analysis of skin filaggrin breakdown products, lipid profiles, and transepidermal water loss will be compared.

SECONDARY OUTCOMES:
Individual reporting of hand dryness and environmental exposures | Through study completion, up to 1 year
  Questionnaires will capture symptoms of hand dryness, frequency of hand washing, and other environmental exposures. This data will be compared to the degree of transepidermal water loss and skin barrier findings.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Hui, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No